CLINICAL TRIAL: NCT01488474
Title: Influence of Diabetic Neuropathy on Current Settings During Peripheral Nerve Stimulation in Regional Anesthesia
Brief Title: Peripheral Nerve Stimulation in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Rigaud Marcel, MD, Principal Investigator, Medical University of Graz
Other Study IDs: KLI 135
Record Dates: First submitted 2011-12-02; First posted 2011-12-08 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Diabetic Polyneuropathy
Keywords: regional anesthesia; peripheral nerve stimulation; diabetes; diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * blood samples
  * any material from surgical resections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes Mellitus (DM): Patients with diagnosed diabetes mellitus type 1 or 2 undergoing surgery of the lower limb and are receiving regional anesthesia with peripheral nerve stimulation
  Interventions: Procedure: peripheral nerve stimulation
- Control (C): Patients with no history of diabetes mellitus Type 1 or 2 undergoing surgery of the lower limb and are receiving regional anesthesia with peripheral nerve stimulation
  Interventions: Procedure: peripheral nerve stimulation

INTERVENTIONS:
Procedure: peripheral nerve stimulation — defining the minimal current threshold for distal motor response

SUMMARY:
The prevalence of diabetes mellitus (DM) in industrialized countries is estimated to be about 7.3% and its incidence has been growing in recent years. The prevalence of diabetic neuropathy in the diabetic patient population is up to 50%. When limb surgery is necessary, it is reasonable to assume that diabetic patients will benefit from a peripheral regional anesthesia because of the severe comorbidities associated with DM. On the other hand, the use of regional anesthesia (RA) has generally not been recommended in patients with preexisting neuropathies mainly because of medical liability issues, as worsening neuropathy could be attributed to nerve damage caused by the regional anesthetic. The current state of the art of peripheral regional anesthesia for the identification of correct placement of an injection needle suitably close to the target nerve is to elicit a motor response by current injection through the needle. Constant reduction of the current as the nerve is approached ensures close proximity so that an effective nerve block is obtained when the local anesthetic is delivered through the needle, and absence of a motor response at 0.3 mA is generally accepted as a safety marker to avoid harmful intraneural injection. An important deficit in our understanding is whether diabetic neuropathy influences the stimulation parameters for peripheral nerve stimulation (PNS), possibly decreasing safety.

The currently proposed research is guided by the hypothesis that nerves in patients with DM are more resistant to stimulation and the current thresholds for PNS have to be set much higher to prevent injections from occurring within the epineurium. The investigators will examine the effect of DM on nerve excitability in a blinded, prospective, observational case control trial. Accordingly, the investigators have defined following aims:

Specific Aim 1: To characterize the required stimulation current in patients with and without diabetes mellitus.

Specific Aim 2: Follow-up to examine if the rate of adverse neurologic events is higher in diabetic patients.

Specific Aim 3: Guided by the results, formulate recommendations for the performance of regional anesthesia in patients with a history of DM.

These experiments will provide better understanding of the needle-current-nerve relationship during peripheral nerve stimulation. Findings from this study will have a major impact on patient safety, especially in the subgroup with preexisting neuropathy, undergoing regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* age more than 18 years
* American Society of Anesthesiology status 1 to 4
* signed informed consent

Exclusion Criteria:

* Pregnancy
* Allergies to local anesthetics
* Unwillingness or incapability to sign informed consent
* Any preexisting neurological deficit of the lower limb that cannot be attributed to diabetic neuropathy
* Ongoing dual anti-platelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients scheduled for lower limb surgery and are eligible for a popliteal sciatic nerve block
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Minimal current threshold for distal motor response at needle tip nerve contact | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Rigaud, PD, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Heschl S, Hallmann B, Zilke T, Gemes G, Schoerghuber M, Auer-Grumbach M, Quehenberger F, Lirk P, Hogan Q, Rigaud M. Diabetic neuropathy increases stimulation threshold during popliteal sciatic nerve block. Br J Anaesth. 2016 Apr;116(4):538-45. doi: 10.1093/bja/aew027. PMID 26994231